CLINICAL TRIAL: NCT04613284
Title: Rh-Endostatin Combined With Low-dose CCRT(50 Gy) Followed by Durvalumab Maintenance for the Treatment of Specific Phase III NSCLC Who Can Not Tolerate 60 Gy Irradiation
Brief Title: Rh-Endostatin Combined With CCRT(50 Gy) Followed by Durvalumab Maintenance for the Treatment of Specific Phase III NSCLC
Acronym: RELIEF
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Chest Hospital (Other)
Collaborators: Wuhan University (Other)
Responsible Party: Principal Investigator, Xuwei Cai, Deputy Chief Physician, Shanghai Chest Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CXW001
Record Dates: First submitted 2020-08-18; First posted 2020-11-03 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Endostatins; endostar protein; durvalumab; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Endostar combined Radiation (Experimental)
  Interventions: Drug: Recombinant human endostatin (Endostar); Radiation: Thoracic irradiation of 50 Gy with 3DCRT or IMRT

INTERVENTIONS:
Drug: Recombinant human endostatin (Endostar) — Continuous intravenous infusion of endostar (Simcere Pharma- ceutical, Nanjing, China) was made over 120 h before the begin- ning of radiotherapy, and then repeated every two weeks. The dose was 7.5 mg/m2/24 h 120 h, 14 days/cycle. ECG monitoring was performed during the first delivery of endostar.
  Other Names: Durvalumab
Radiation: Thoracic irradiation of 50 Gy with 3DCRT or IMRT — Concurrent thoracic chemoradiotherapy with reduced irradiation dose of 50 Gy will be given to patients with unresectable stage III NSCLC who can not tolerate irradiation dose to 60 Gy.

SUMMARY:
A Study to Assess the Effects of Durvalumab following Rh-Endostatin combined with reduced-dose CCRT(50 Gy) in Patients with Stage III Unresectable Non-Small Cell Lung Cancer who can not tolerate 60 Gy irradiation.

DETAILED DESCRIPTION:
A Phase II, Single-arm, Multi-centre Study of Durvalumab as Sequential Therapy in Patients with Locally Advanced, Unresectable Non-Small Cell Lung Cancer (Stage III) Who Have Not Progressed Following Rh-Endostatin combined with reduced-dose CCRT(50 Gy) Therapy (Relief)

ELIGIBILITY:
Inclusion Criteria:

* Age at 18-75 years.
* Documented evidence of NSCLC (locally advanced, unresectable, Stage III)
* Measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST)
* Eastern Cooperative Oncology Group performance status score (ECOG PS) of 0 to 1.
* Estimated life expectancy of more than 12 weeks.

Exclusion Criteria:

* Prior exposure to any anti-PD-1 or anti-PD-L1 antibody.
* Active or prior autoimmune disease or history of immunodeficiency.
* Evidence of severe or uncontrolled systemic diseases, including active bleeding diatheses or active infections including hepatitis B, C and HIV.
* Evidence of uncontrolled illness such as symptomatic congestive heart failure, uncontrolled hypertension or unstable angina pectoris.
* Any unresolved toxicity CTCAE >Grade 2 from the prior chemoradiation therapy.
* Active or prior documented inflammatory bowel disease (eg, Crohn's disease, ulcerative colitis).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2022-02 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | up to approximately 3 years
  PFS was defined as the time from randomization until the date of objective disease progression (RECIST 1.1) or death (by any cause in the absence of progression).
adverse events (AE) | 5 years from patient enrollment
  Number of participants with adverse events as assessed by CTCAE v5.0

SECONDARY OUTCOMES:
Overall Survival | up to 5 years from patient enrollment
  OS was defined as the time from the date of randomization until death due to any cause. OS was calculated using the Kaplan-Meier technique.
Objective Response Rate | Tumor scans performed at baseline then every ~8 weeks up to 48 weeks, then every ~ 12 weeks thereafter up to 3 three years
  ORR was defined as the percentage of patients with at least one visit response of Complete Response (CR) or Partial Response (PR) per RECIST 1.1 for target lesions: CR: Disappearance of all target lesions; PR: >=30% decrease in the sum of the longest diameter of target lesions; OR = CR + PR.